CLINICAL TRIAL: NCT04987671
Title: A Pharmacokinetic and Pharmacodynamic Study of AMX0035 in Patients With ALS
Brief Title: Pharmacokinetic and Pharmacodynamic Study of AMX0035 in Patients With ALS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A35-005
Record Dates: First submitted 2021-07-15; First posted 2021-08-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: ALS
Keywords: Neurodegenerative Diseases; Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Nervous System Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Neurodegenerative Diseases; Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Nervous System Diseases; Neuromuscular Diseases | interventions — sodium phenylbutyrate and taurursodiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with AMX0035 (Experimental): Two sequential study period. In Period 1, subject receive AMX0035 daily for approximately 14 days. In Period 2, subjects receive AMX0035 twice a day, morning and evening, for up to 25 days.
  Interventions: Drug: AMX0035

INTERVENTIONS:
Drug: AMX0035 — Fixed dose combination of Sodium Phenylbutyrate and taurursodiol.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic and pharmacodynamic effect after a single dose or at steady state after multiple doses of AMX0035 in adults with sporadic ALS.

DETAILED DESCRIPTION:
AMX0035 is a proprietary combination of two small molecules, phenylbutyrate (PB) and taurursodiol. The combination of PB and taurursodiol in AMX0035 is intended to block neuronal death and neurotoxic inflammation through simultaneous reduction of endoplasmic reticulum (ER) stress and mitochondrial stress. The pharmacokinetic of AMX0035 has been evaluated in healthy volunteers. This Phase IIa trial is intended to evaluate pharmacokinetic of PB and taurursodiol upon single dose multiple dose administration of AMX0035 in patients with ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >=18years of age;
2. Diagnosis of sporadic ALS (definite, probable, laboratory probable, possible) made by physician experienced with management of ALS as defined by the World Federation of Neurology revised El Escorial criteria;
3. If taking riluzole, must be on a stable dose for >30 days prior to Day 1 and anticipated to remain at that dose until the final study visit.
4. If taking edaravone, must be on a stable regimen for > 30 days prior to Day 1 and infusion(s) can be scheduled to be performed at no less than 48 hours prior or after the planned pharmacokinetic and pharmacodynamic (PK/PD) sampling.
5. Capable of providing informed consent and following trial procedures;
6. Geographically accessible to the site;
7. Able to undergo the study procedures (including planned sampling on 3 occasions) and to adhere to the visit schedule, as determined by Investigator;
8. Women of child bearing potential (e.g. not post-menopausal for at least one year or surgically sterile) must agree to use adequate birth control for the duration of the study and 3 months after last dose of study drug;

   a. Women must not be planning to become pregnant for the duration of the study and 3 months after last dose of study drug
9. Men must agree to practice contraception for the duration of the study and for at least 3 months after last dose of study drug;

   1. Men must not plan to father a child or provide sperm for donation for the duration of the study and 3 months after last dose of study drug
   2. Acceptable birth control methods for use in this study are:

      * Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
      * Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
      * Intrauterine device (IUD)
      * Abstinence (no heterosexual sex)
      * Unique partner who is surgically sterile (men) or not of child bearing potential (female)

Exclusion Criteria:

1. Familial ALS
2. Forced vital capacity < 50% (or alternatively SVC) or presence of tracheostomy or under PAV (PAV is defined as more than 22 hours daily of non-invasive mechanical ventilation for more than 7 days);
3. Planned elective surgery (such as feeding tube or edaravone access port placement) during the duration of the study;
4. History of known allergy to PB or bile salts;
5. Abnormal liver function defined as aspartate aminotransferase and/or alanine aminotransferase (AST and/or ALT) > 3 times the upper limit of the normal;
6. Renal insufficiency as defined by eGFR < 60 mL/min/1.73m2;
7. Ongoing Anemia with Hg concentration < 10.0 g/dL
8. Pregnant women or women currently breastfeeding;
9. Current biliary disease which may lead to biliary obstruction or impedes biliary flow including active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gallbladder polyps, gangrene of the gallbladder, abscess of the gallbladder;
10. History of Class III/IV heart failure (per New York Heart Association - NYHA);
11. Patient under severe salt restriction where the added salt intake due to treatment would put the patient at risk, in the Site Investigator clinical judgement;
12. Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the subject to provide informed consent, according to Site Investigator judgment;
13. Presence of an active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period.
14. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the subject if they were to participate in the study, according to Site Investigator judgment.
15. Clinically significant, as determined by the Investigator, 12-lead ECG abnormalities at screening.
16. Treatment, current or within 90 days from start of study treatment, with any cell therapies or gene therapies;
17. Treatment, current or within 90 days from start of study treatment, with experimental medication (for ALS or other indications)
18. Current or anticipated need for a Diaphragm Pacing System (DPS);
19. Anything that, in the opinion of the Site Investigator preclude the subject's full compliance with or completion of the study;
20. Exposure to any disallowed medications listed below:

    1. HDAC Inhibitors including:

       * Valproate
       * Vorinostat (Zolinza)
       * Romidepsin
       * Chidamide
       * Panobinostat
       * Lithium
       * Butyrate
       * Suramin
    2. Probenecid
    3. Bile Acid Sequestrants including:

       * Cholestyramine and Cholestyramine Light
       * Questran and Questran Light
       * Welchol
       * Colestid and Colestid Flavored
       * Prevalite
    4. Product that may interact with sterol absorption or excretion

       * Ezetimibe
    5. Note on Antacids within Two Hours of AMX0035 Administration: Antacids containing aluminum hydroxide or smectite (aluminum oxide) may not be taken within two hours of administration of MX0035 as they inhibit absorption of taurursodiol. These include:

       * Alamag
       * Alumina and Magnesia
       * Antacid, Antacid M and Antacid Suspension
       * Gen-Alox
       * Kudrox
       * M.A.H.
       * Maalox HRF and Maalox TC
       * Magnalox
       * Maldroxal
       * Mylanta and Mylanta Ultimate
       * Ri-Mox
       * Rulox
21. Clinically significant, in the opinion of the Investigator, infection or inflammation at time of screening or admission.
22. Acute gastrointestinal symptoms (eg, nausea, vomiting, diarrhea) at time of screening or admission or a or clinical diagnosis of irritable bowel syndrome (IBS) per ROME criteria (Appendix 7).
23. Any current or previous illicit use of Class A drugs such as opiates, cocaine, ecstasy, LSD, and amphetamines (Class B).
24. An alcoholic intake greater than 14 units per week or unwillingness to stop alcohol consumption for the duration of the study. Note: 1 unit = 8 g ethanol (250 mL of beer or approximately 10 oz, 1 glass wine [100 mL or approximately 3 oz], 1 measure spirits [30 mL or approximately 1 oz]).
25. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of investigational product.
26. History of plasma/blood donation in the last 2 months.
27. Any condition, which compromises ability to give informed consent or to communicate with the Investigator as required for the completion of this study.
28. Unwilling to conform to all lifestyle considerations and restrictions mandated by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Blood concentration of PB and taurursodiol | Between Day 1 and Day 40
  Maximum plasma concentration - Cmax of PB and taurursodiol
Systemic exposure to PB and taurursodiol | Between Day 1 and Day 40
  Area under the plasma concentration versus time curve - AUC of PB and taurursodiol

SECONDARY OUTCOMES:
Effect of demographic characteristics on blood concentration of PB and taurursodiol | Between Day 1 and Day 40
  Maximum plasma concentration - Cmax of PB and taurursodiolin relation to gender, body weight and age.
Effect of demographic characteristics on systemic exposure of PB and taurursodiol | Between Day 1 and Day 40
  Area under the plasma concentration versus time curve - AUC of PB and taurursodiol relation to gender, body weight and age.
Effect of a fixed dose combination of sodium phenyl butyrate (PB) and taurursodiol on pharmacodynamic activity | Between Day 1 and Day 40
  Histone 3 and histone 4 acetylation levels in peripehral blood mononuclear cells (PBMC)

CONTACTS AND LOCATIONS:
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuadrado-Tejedor M, Ricobaraza AL, Torrijo R, Franco R, Garcia-Osta A. Phenylbutyrate is a multifaceted drug that exerts neuroprotective effects and reverses the Alzheimer s disease-like phenotype of a commonly used mouse model. Curr Pharm Des. 2013;19(28):5076-84. doi: 10.2174/1381612811319280006. PMID 23448463
- [Background] Cudkowicz ME, Andres PL, Macdonald SA, Bedlack RS, Choudry R, Brown RH Jr, Zhang H, Schoenfeld DA, Shefner J, Matson S, Matson WR, Ferrante RJ; Northeast ALS and National VA ALS Research Consortiums. Phase 2 study of sodium phenylbutyrate in ALS. Amyotroph Lateral Scler. 2009 Apr;10(2):99-106. doi: 10.1080/17482960802320487. PMID 18688762
- [Background] Nunes AF, Amaral JD, Lo AC, Fonseca MB, Viana RJ, Callaerts-Vegh Z, D'Hooge R, Rodrigues CM. TUDCA, a bile acid, attenuates amyloid precursor protein processing and amyloid-beta deposition in APP/PS1 mice. Mol Neurobiol. 2012 Jun;45(3):440-54. doi: 10.1007/s12035-012-8256-y. Epub 2012 Mar 23. PMID 22438081
- [Background] Dionisio PA, Amaral JD, Ribeiro MF, Lo AC, D'Hooge R, Rodrigues CM. Amyloid-beta pathology is attenuated by tauroursodeoxycholic acid treatment in APP/PS1 mice after disease onset. Neurobiol Aging. 2015 Jan;36(1):228-40. doi: 10.1016/j.neurobiolaging.2014.08.034. Epub 2014 Sep 28. PMID 25443293
- [Background] Lo AC, Callaerts-Vegh Z, Nunes AF, Rodrigues CM, D'Hooge R. Tauroursodeoxycholic acid (TUDCA) supplementation prevents cognitive impairment and amyloid deposition in APP/PS1 mice. Neurobiol Dis. 2013 Feb;50:21-9. doi: 10.1016/j.nbd.2012.09.003. Epub 2012 Sep 10. PMID 22974733
- [Background] Ricobaraza A, Cuadrado-Tejedor M, Marco S, Perez-Otano I, Garcia-Osta A. Phenylbutyrate rescues dendritic spine loss associated with memory deficits in a mouse model of Alzheimer disease. Hippocampus. 2012 May;22(5):1040-50. doi: 10.1002/hipo.20883. Epub 2010 Nov 10. PMID 21069780
- [Background] Ricobaraza A, Cuadrado-Tejedor M, Perez-Mediavilla A, Frechilla D, Del Rio J, Garcia-Osta A. Phenylbutyrate ameliorates cognitive deficit and reduces tau pathology in an Alzheimer's disease mouse model. Neuropsychopharmacology. 2009 Jun;34(7):1721-32. doi: 10.1038/npp.2008.229. Epub 2009 Jan 14. PMID 19145227
- [Background] Rodrigues CM, Sola S, Sharpe JC, Moura JJ, Steer CJ. Tauroursodeoxycholic acid prevents Bax-induced membrane perturbation and cytochrome C release in isolated mitochondria. Biochemistry. 2003 Mar 18;42(10):3070-80. doi: 10.1021/bi026979d. PMID 12627974
- [Background] Wiley JC, Pettan-Brewer C, Ladiges WC. Phenylbutyric acid reduces amyloid plaques and rescues cognitive behavior in AD transgenic mice. Aging Cell. 2011 Jun;10(3):418-28. doi: 10.1111/j.1474-9726.2011.00680.x. Epub 2011 Mar 22. PMID 21272191
- [Background] Wright JM, Zeitlin PL, Cebotaru L, Guggino SE, Guggino WB. Gene expression profile analysis of 4-phenylbutyrate treatment of IB3-1 bronchial epithelial cell line demonstrates a major influence on heat-shock proteins. Physiol Genomics. 2004 Jan 15;16(2):204-11. doi: 10.1152/physiolgenomics.00160.2003. PMID 14583596
- [Background] Zhou W, Bercury K, Cummiskey J, Luong N, Lebin J, Freed CR. Phenylbutyrate up-regulates the DJ-1 protein and protects neurons in cell culture and in animal models of Parkinson disease. J Biol Chem. 2011 Apr 29;286(17):14941-51. doi: 10.1074/jbc.M110.211029. Epub 2011 Mar 3. PMID 21372141